CLINICAL TRIAL: NCT05540275
Title: Phase 2 Study to Evaluate the Clinical Efficacy and Safety of Tislelizumab Plus Low-dose Bevacizumab in Bevacizumab Refractory Recurrent Glioblastoma With PTEN or TERT Gene Mutations
Brief Title: Tislelizumab (One Anti-PD-1 Antibody) Plus Low-dose Bevacizumab for Bevacizumab Refractory Recurrent Glioblastoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HenanPPH-Recurrent GBM
Record Dates: First submitted 2022-09-11; First posted 2022-09-14 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — tislelizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Patients with bevacizumab-refractory recurrent glioma with PTEN or TERT gene mutations,determined according to the dynamics of TISF (Tumor in Situ Fluid) ctDNA.
  Interventions: Drug: Tislelizumab plus Bevacizumab
- Cohort 2 (Experimental): Patients with bevacizumab-refractory recurrent glioma without PTEN or TERT gene mutations,determined according to the dynamics of TISF (Tumor in Situ Fluid) ctDNA.
  Interventions: Drug: Tislelizumab plus Bevacizumab

INTERVENTIONS:
Drug: Tislelizumab plus Bevacizumab — 200mg Tislelizumab plus 3mg/kg bevacizumab every 3 weeks

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety of Tislelizumab (one anti-PD-1 antibody same as nivolumab approved in China) in combination with bevacizumab in patients with recurrent or progressive glioblastoma (GBM) who have progressed on bevacizumab with or without PTEN or TERT gene mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations
2. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of thestudy, including disease assessment by MRI and tumor in situ fluid (TISF) collection
3. Histologically confirmed diagnosis of glioma
4. Resection surgery done at the study center (Henan Provincial People'sHospital), with an reservoir intraoperatively implanted connecting the surgical cavity and the subscalp for postoperative noninvasive TISF collection
5. An interval of > 28 days and full recovery (i.e., no ongoing safety issues) from surgical resection prior to grouping
6. Karnofsky performance status (KPS) of 70 or higher
7. Life expectancy > 12 weeks

Exclusion Criteria:

1. More than two recurrences of GBM
2. Presence of extracranial metastatic, significant leptomeningeal disease or tumors primarily localized to the brainstem or spinal cord
3. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results
4. Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring chronic and systemic immunosuppressive treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll. Subjects have any other condition requiring systemic treatment with corticosteroids or other immunosuppressive agents within 14 days. Inhaled or topical steroids and adrenal replacement doses >10mg daily prednisone equivalent are permitted in absence of active autoimmune disease
5. Previous radiation therapy with anything other than standard radiation therapy (i.e., focally directed radiation) administered as first line therapy
6. Previous treatment with carmustine wafer except when administered as first line treatment and at least 6 months prior to randomization
7. Previous bevacizumab or other VEGF or anti-angiogenic treatment
8. Previous treatment with a PD-1, PD-L1 or CTLA-4 targeted therapy
9. Evidence of > Grade 1 CNS hemorrhage on the baseline MRI scan
10. Inadequately controlled hypertension (defined as systolic blood pressure ≥160 mmHg and /or diastolic blood pressure ≥100 mmHg) within 7 days of first study treatment
11. Prior history of hypertensive crisis, hypertensive encephalopathy, reversible posterior leukoencephalopathy syndrome (RPLS)
12. Prior history of gastrointestinal diverticulitis, perforation, or abscess
13. Clinically significant (i.e., active) cardiovascular disease, for example cerebrovascular accidents ≤ 6 months prior to study enrollment, myocardial infarction ≤ 6 months prior to study enrollment, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure (CHF), or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with protocol treatment
14. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to start of study treatment. Any previous venous thromboembolism ≥ NCI CTCAE Grade 3 within 3 months prior to start of study treatment
15. History of pulmonary hemorrhage/hemoptysis ≥ grade 2 (defined as ≥ 2.5 mL bright red blood per episode) within 1 month prior to randomization
16. History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e., in the absence of therapeutic anticoagulation)
17. Current or recent (within 10 days of study enrollment) use of anticoagulants that, in the opinion of the investigator, would place the subject at significant risk for bleeding. Prophylactic use of anticoagulants is allowed
18. Surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to first study treatment, or anticipation of need for major surgical procedure during the course of the study
19. Minor surgical procedure (e.g., stereotactic biopsy within 7 days of first study treatment; placement of a vascular access device within 2 days of first study treatment)
20. History of intracranial abscess within 6 months prior to randomization
21. History of active gastrointestinal bleeding within 6 months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to 2 years after beginning treatment
  Proportion of participants in the analysis population who have complete response (CR) or partial response (PR) using RANO criteria. Participants without efficacy evalaluation data or survival data censored at day 1. Participants without measurable disease will not be included.
Duration of response | Up to 2 years after beginning treatment
  Time from first RANO response to disease progression in participants who achieve a PR or better.
Number of participants with treatment-emergent adverse events | Up to 3 months after beginning therapy
  Toxicity is graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. Adverse events (AEs) are reported based on clinical laboratory tests, vital sign and weight measurements, physical examinations, performance status evaluations, magnetic resonance imaging, and any other medically indicated assessments, including subject interviews, from the time informed consent is signed through 90 days after the last dose of durvalumab. AEs are considered to be treatment emergent if they occur or worsen in severity after the first dose of study treatment.

SECONDARY OUTCOMES:
Overall survival | Up to 2 years after beginning treatment
  overall survival, as defined as time from beginning of treatment to death.

CONTACTS AND LOCATIONS:
Overall Officials: Xingyao Bu, MD, PhD, Study Director — Henan Provincial People's Hospita
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo G, Zhang Z, Zhang J, Wang D, Xu S, Liu G, Gao Y, Mei J, Yan Z, Zhao R, Wang M, Li T, Bu X. Predicting recurrent glioblastoma clinical outcome to immune checkpoint inhibition and low-dose bevacizumab with tumor in situ fluid circulating tumor DNA analysis. Cancer Immunol Immunother. 2024 Aug 6;73(10):193. doi: 10.1007/s00262-024-03774-7. PMID 39105794